CLINICAL TRIAL: NCT06022874
Title: The Therapeutic Effects of Topical Cannabidiol (CBD) Products for Atopic Dermatitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Phoilex Ltd. (Industry)
Collaborators: Phoenix Medical Spa X Peak Human (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00066042
Record Dates: First submitted 2023-08-28; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient's Diagnosed with Atopic Dermatitis: Patient's Diagnosed with Atopic Dermatitis
  Interventions: Other: Phoilex Releaf Gel

INTERVENTIONS:
Other: Phoilex Releaf Gel — Patients will be given the Releaf Gel to apply to the affected areas daily. They will be examined at the following time points: Immediately after application, 1 week, 2 weeks, and 4 weeks.
  The instructions given to the patient shall be to apply one pump per every affected area, wash hands before applying to affected area, apply twice a day (morning, and evening), apply on clean skin, and application after showering is advised.
  The number of pumps of Phoilex Releaf gel will be documented within a chart provided to the patient. It is suggested that not more than 25 lesions compassing an area greater than 50 cm² in total be treated during the course of this study.
  The maximum dose would be 240 mL of Phoilex Releaf gel in 30 days. The minimum dose would be 0.5 mL (one pump) of the Phoilex Releaf gel in 30 days. The maximum daily dose of CBD per day 46 mg per application, equivalent to 92 mg per day.

SUMMARY:
The goal of this observational study is to learn about the potential therapeutic effects of topical CBD products produced by Phoilex Ltd., specifically the Releaf Gel, in those diagnosed with atopic dermatitis. Patients will be routinely assessed via questionnaire, and physical measurements will be taken with respect to the affected area studied in order to judge clinical efficacy.

The main question[s] it aims to answer are:

* Did you experience an immediate increase in skin hydration?
* Did you experience a soothing or comforting feeling on your irritated skin area? Please explain where your affected area is located, and also include at what time point this occurred. Example: Affected Area: Palm, Time Point: 1-hour post-application
* Upon the affected area being in the healing phase, was your skin itch/scratch free for 4/6/10/12 hours (please circle)?
* Did you experience immediate relief from your skin inflammation?
* Did the study cream absorb quickly into your skin, without any greasy feeling?
* Has your skin flare disappeared in 2 week(s)?
* Has your skin condition appearance improved? (Yes/No)

Participants will apply Phoilex Releaf Gel (a cream) to their affected areas of atopic dermatitis. The questions listed above shall be discussed and observations recorded at the 0 week, 1 week, 2 week, and 4 week time points. Additional monitoring questions may be asked of the participants to ensure the safety of the product. A chart will be provided to the participants to track Phoilex Releaf Gel usage (how many pumps, and time of day) throughout duration of the study.

We hypothesize that Releaf gel will be suitable to ameliorate the common signs and symptoms of atopic dermatitis as well as improve patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Specifically, patients would be recruited based on the following inclusion criteria must be over 18 years old and must be diagnosed with moderate-to-severe eczema.

Exclusion Criteria:

* Exclusion criteria would include not currently using any steroids or biologics, not currently using any other topical products, not pregnant, not breast feeding, nor have any allergies to any ingredients listed within the formula of the Releaf gel. A negative pregnancy test will need to be confirmed prior to patient receiving Phoilex Releaf Gel. Lastly, participants who have been diagnosed with anxiety or depression with a classification of greater than mild anxiety or mild depression will be excluded. As such, screening for possible candidates for the clinical trial will include questions and a brief assessment on participants mental health by study doctor/physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with moderate to severe atopic dermatitis will be selected and recruited from medical clinics, social media, as well as invitation should they meet the inclusion criteria. Participants must be able to travel to clinic location in Brampton.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Will topically applied CBD be effective in reducing the appearance/clearing of atopic dermatitis after 4 weeks of study treatment? | 5 weeks
  Outcome will be measured based on observations recorded at 0 weeks, 1 week, 2 week, and 4 week time point, not limited to physical assessment, clinical photography, and the responses of questions below:
  * Did you experience an immediate increase in skin hydration?
  * Did you experience a soothing or comforting feeling on your irritated skin area? Please explain where your affected area is located, and also include at what time point this occurred. Example: Affected Area: Palm, Time Point: 1-hour post-application
  * Upon the affected area being in the healing phase, was your skin itch/scratch free for 4/6/10/12 hours (please circle)?
  * Did you experience immediate relief from your skin inflammation?
  * Did the study cream absorb quickly into your skin, without any greasy feeling?
  * Has your skin flare disappeared in 2 week(s)?
  * Has your skin condition appearance improved? (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Goel, MD, Principal Investigator — Phoenix Medical Spa X Peak Human
Locations (1):
- Phoenix Medical Spa X Peak Human, Brampton, Ontario, Canada